CLINICAL TRIAL: NCT02341651
Title: Feasibility Study for a Cluster Randomized Trial on Integrated Primary Care Strategies to Reduce High Blood Pressure (Control of Blood Pressure and Risk Attenuation-rural Bangladesh, Pakistan, Sri Lanka, Feasibility Study)
Brief Title: Control of Blood Pressure and Risk Attenuation-rural Bangladesh, Pakistan, Sri Lanka, Feasibility Study
Acronym: COBRA-BPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Aga Khan University (Other); University of Kelaniya (Other)
Responsible Party: Principal Investigator, Professor Tazeen Jafar, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MR/L004224/1
Record Dates: First submitted 2014-12-28; First posted 2015-01-19 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: High blood pressure; Cardiovascular diseases; Antihypertensive agents; Pharmacological treatment; Non-pharmacological treatment; Community health care workers; Treatment algorithm; Public and private healthcare providers; Strategy; Referral loops; Intervention
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multicomponent "combination" (Experimental): Multicomponent intervention is a combination of the following 1) community health worker (CHW)- led blood pressure (BP) screening and referral to provider, plus 2) home health education (HHE) adapted to the local diet by trained CHW plus 3) trained primary health center mid-level providers (MLP) and physicians using evidence-based treatment algorithm of BP lowering in all and lipid lowering for high risk, plus 4) process-based incentives
  Interventions: Other: Multicomponent intervention
- Usual Care (No Intervention): No active intervention

INTERVENTIONS:
Other: Multicomponent intervention — Multicomponent intervention is a combination of the following 1) community health worker (CHW)- led blood pressure (BP) screening and referral to provider, plus 2) home health education (HHE) adapted to the local diet by trained CHW plus 3) trained primary health center mid-level providers (MLP) and physicians using evidence-based treatment algorithm of BP lowering in all and lipid lowering for high risk, plus 4) process-based incentives
  Arms: Multicomponent "combination"

SUMMARY:
High blood pressure (BP) is the leading attributable risk for cardiovascular disease (CVD). In rural South Asia, hypertension remains to be a significant public health issue with sub-optimal rates of case finding and management. A trial to investigate integrated primary care strategies to control hypertension is planned. Packaged interventions for the planned full-scale study are varying combinations of 1) home health education (HHE) by trained community health workers (CHW), 2) trained government primary health centre mid-level providers (MLP) led care and 3) trained private practitioners. The goal of the full-scale study is to test which combination of the above interventions is the most effective in lowering blood pressure among adults with hypertension in rural communities. In addition, the full-scale study aims to quantify the incremental cost- effectiveness of each approach in terms of cost per projected cardiovascular disease (CVD) disability adjusted life-years (DALYs) averted.

DETAILED DESCRIPTION:
The rationale for conducting the feasibility study in 3 proposed South Asian countries is strong. The South Asian countries are in a unique stage of epidemiological transition with a double burden of communicable and NCDs, the latter increasing rapidly. (2) These countries also share cultural habits and social structure with an extended family system, and have largely similar population characteristics and health seeking behaviours. (10)Moreover, the rural health system in all South Asian countries relies on cadres community health workers. At the same time there are some differences. Bangladesh and Pakistan have a high proportion of people living in extreme poverty (purchasing power parity <US $1.25/day, 49.6% and 22.6%, respectively) compared to Sri Lanka (14%) which has relatively better development indicators in terms of life expectancy and literacy rates (World Bank 2010). However age-standardized death rates from non-communicable diseases (NCDs) are uniformly high in all 3 countries. The feasibility will allow direct comparison of some of these population (individual) and health systems characteristics among countries relevant for hypertension care. Thus, data from the feasibility will inform the future design of the trial.

In order to optimize the trial design of the full study, a mixed-methods feasibility study with quasi-experimental pre- and post- evaluation of "triple approach" with all 3 components of intervention, survey of pharmacies, and focus group discussions and individual in-depth interviews to better inform the strategies for the full-scale trial in rural settings in Bangladesh, Pakistan, and Sri Lanka.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 40 years
2. Residing in the selected clusters
3. Hypertension defined either as:

   1. persistently elevated BP (systolic BP ≥140 mm Hg or diastolic BP ≥90 mm Hg) from each set of 2 readings from 2 separate days
   2. maintained on anti-hypertensive medications
4. Informed consent

Exclusion Criteria:

1. Bed-ridden individuals too ill to commute to the clinic
2. Individuals with advanced medical disease (on dialysis, liver failure, other systemic diseases)
3. Individuals that are mentally compromised and unable to give informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
retention rate | 3 months
  proportion of hypertensive individuals followed up at 3 months in 3 countries

SECONDARY OUTCOMES:
Fidelity measure- Proportion of providers trained | 3 months
  proportion of targeted providers trained in 3 countries
Fidelity measure- home health education sessions delivered | 3 months
  Proportion of planned home health education sessions delivered in 3 countries
fidelity measure 3- physician management checklist collected | 3 months
  proportion of expected physician management checklist collected
Baseline to follow-up change in systolic blood pressure level | 3 months
  within clusters intra-class correlation (95% CI) pre- to post- intervention change in systolic

CONTACTS AND LOCATIONS:
Overall Officials: Tazeen H Jafar, MD, MPH, Principal Investigator — Duke-NUS, Singapore; Aliya Naheed, Principal Investigator — Initiative for Non-Communicable Diseases icddr,b, Bangladesh; Imtiaz Jehan, Principal Investigator — Aga Khan University; Asita de Silva, Principal Investigator — University of Kelaniya, Sri Lanka; Shah Ebrahim, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (3):
- Initiative for Non-Communicable Diseases icddr,b, Dhaka, Mohakhali, Bangladesh
- Aga Khan University Hospital, Karachi, Karachi, Pakistan
- University of Kelaniya, Ragama, Ragama, Sri Lanka

REFERENCES:
- [Derived] Jafar TH, Silva Ad, Naheed A, Jehan I, Liang F, Assam PN, Legido-Quigley H, Finkelstein EA, Ebrahim S, Wickremasinghe R, Alam D, Khan AH; COBRA-BPS Study Group. Control of blood pressure and risk attenuation: a public health intervention in rural Bangladesh, Pakistan, and Sri Lanka: feasibility trial results. J Hypertens. 2016 Sep;34(9):1872-81. doi: 10.1097/HJH.0000000000001014. PMID 27488552